CLINICAL TRIAL: NCT02895399
Title: Epidémiologie de l'Infection à Human Papilloma Virus Chez Les Femmes Vivant Sur Les Fleuves Maroni et Oyapock
Brief Title: Epidemiology of Human Papillomavirus Infection Among Women Living on the Maroni and the Oyapock Rivers
Acronym: EPHaVI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: 30814
Record Dates: First submitted 2016-09-05; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Human Papillomavirus Viruses

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cervico-Vaginal Smears
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Cervico-Vaginal Smears analysis — Cervico-Vaginal Smears analysis

SUMMARY:
Cervical cancer is the second most frequent cancer of women in French Guiana. Studies have shown that populations living in remote villages in the interior of the territory have early sexual relations and that multiple sexual partnerships are frequent. Hence, the main objective of the study was to determine the prevalence of HPV in these areas, and the predictive factors and epidemiology of this viral infection.

Methods - This multicentric cross sectional study aimed the population of women aged 20 to 65 years, living in the remote villages along the Maroni and Oyapock rivers. Women wishing to participate will be included after being informed of the study team schedule through radio address and key opinion leaders. The search for HPV and cytologic examinations will be performed for each woman. 2 samples will be taken from each woman: one sample will be sent to Fort De France hospital for cytology, and HPV testing; cytologic analyses will be performed using the 2001 Bethesda classification. Another sample will be sent to Pasteur Institute in Cayenne for sequencing and detection of E6 and E7 RNA which are associated with carcinogenesis. HPV infection will be defined by the detection of viral DNA using the GREINER-BIO-ONE kit. Statistical analysis of the results will use STATA software and mapping will use Mapinfo.

ELIGIBILITY:
Inclusion Criteria:

* Women aged from 20 to 65 living in a common Maroni rivers (Apatou , Grand Santi, Papaichton , Maripasoula and the Native American territory of Upper Maroni) and / or Oyapock ( Saint Georges, Camopi , Three Jumps )
* Having already had sexual intercourse
* Having given after information , consent to the inclusion in the study

Exclusion Criteria:

* Age < 20 or age> 65 years
* Being pregnant more than 3 months
* Have had a hysterectomy
* Denial of participation

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: women from 20 to 65 years living on the Maroni and the Oyapock rivers having already had sexual intercourse
Sampling Method: Non-Probability Sample
Enrollment: 643 (Actual)
Dates: Start 2012-12; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Prevalence and distribution of Human Papillomaviruses genotypes | At the time of inclusion (baseline)